## Postcard Consent -

**Protocol #: 21-4768** 

Project Title: Health system methods to improve nursing retention amidst ongoing

COVID-19 pandemic: a mixed-method study

Study Title: HEALTH SYSTEM METHODS TO IMPROVE NURSING RETENTION AMIDST

ONGOING COVID-19 PANDEMIC: A MIXED-METHOD STUDY

Principal Investigator: Claire Aksamit, PA-C; Lacey LaGrone, MD; Laura Ellis, RN

**COMIRB No: 21-4768** 

Version #: 2

Version Date: February 10, 2022

You are being asked to participate in this research study because you currently are or were recently employed as an administrative or clinical staff member of UCHealth Medical Center of the Rockies on the Trauma/Surgical floor or Surgical ICU in the last 24 months. Our research team is enrolling participants like you to identify barriers and facilitators to hospital nursing retention.

If you join the study, you will be asked to complete a confidential in-person or virtual interview with the trained study team that will last approximately 30-45 minutes. The interview will be recorded on a digital recorder and then transcribed. All data will be kept in encrypted files and only accessed by the core research team. All transcripts will be destroyed within five years after the study concludes in compliance with FDA requirements. At the end of the survey, you may be asked to share the study with prior nurse employees who have left the Trauma/Surgical floor, SPCU, or Surgical ICU at Medical Center of the Rockies in the past approximately 24 months who may be interested in participating and be given our contact information to pass along to them. In addition, there will be a four-question survey that will take approximately two minutes that will be sent via email at a later time

This study is designed to learn more about the emotional and physical stress, worsening compassion fatigue, and burnout of nurses as a result of the coronavirus pandemic. Global healthcare systems continue to lose nurses. Administrators and health care systems have implemented additional resources such as financial incentives and emotional support programs to improve provider and staff retention. However, there is an urgency to understand better how hospital systems can improve nursing retention. The purpose of this study is to evaluate different means of improving nursing retention by collecting first-hand accounts from affected employees.

Risks include discomfort in answering interview questions and a possible loss of confidentiality. The interview data will be de-identified to protect the confidentiality of your participation. There may be risks the researchers have not thought of. At any point, you may choose not to answer a question, and the interview may be terminated if you wish.

This study is not designed to benefit you directly.

Every effort will be made to protect your privacy and confidentiality by de-identifying your responses.

You have a choice about being in this study. You do not have to be in this study if you do not want to be. You may leave the study at any time. You will not be paid for taking part in this study. You will not incur any additional costs for participation.

The data we collect will be used for this study but may also be important for future research. Your data may be used for future research or distributed to other researchers for future study without additional consent if information that identifies you is removed from the data.

Study Title: HEALTH SYSTEM METHODS TO IMPROVE NURSING RETENTION AMIDST ONGOING COVID-19 PANDEMIC: A MIXED-METHOD STUDY

Principal Investigator: Claire Aksamit, PA-C; Lacey LaGrone, MD; Laura Ellis, RN

**COMIRB No: 21-4768** 

Version #: 2

Version Date: February 10, 2022

The analysis of the data collected may be shared at meetings and with management at UCHealth. The results of the study may also be included in relevant journals; however, individuals will not be identified.

If you have questions, you can call Claire Aksamit, PA-C at (507) 261-4782 or Lacey LaGrone, MD, at (970) 203-7259 at any time.

You may have questions about your rights as someone in this study. If you have questions, you can call COMIRB (the responsible Institutional Review Board) at (303) 724-1055.

By providing your electronic signature, you are agreeing to participate in this research study.

| Signature: |
|------------|
| Date: |